CLINICAL TRIAL: NCT02976727
Title: Efficacy of Topical Calcipotriol-assisted Ablative Fractional Laser Photodynamic Therapy for the Treatment of Actinic Keratosis: 12-month Follow-up Results of a Prospective, Randomised, Comparative Trial
Brief Title: Efficacy of Topical Calcipotriol-assisted AFL-PDT in Actinic Keratosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A University (Other)
Responsible Party: Principal Investigator, Song Ki-Hoon, Assistant professor and chairman, Department of dermatology Dong-A University, College of medicine, Dong-A University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: DAUderma-07
Record Dates: First submitted 2016-11-05; First posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Actinic Dermatosis
Keywords: Vitamin D; Calcipotriol; Ablative fractional laser; Actinic keratosis; Photodynamic therapy
MeSH Terms: conditions — Keratosis, Actinic | interventions — Vitamin D; calcipotriene; Lidocaine; Prilocaine; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GroupA (Vit-D pretreated AFL-PDT group ) (Experimental): Group A was treated with topical VitD-assisted AFL-PDT
  Interventions: Drug: Topical Vitamin D (Calcipotriol) application; Drug: lidocaine/prilocaine (5%) application; Device: 2940-nm Er:YAG AFL pretreatment; Drug: MAL application; Other: Measurements of the fluorescence intensity; Device: irradiation with red light-emitting diode lamp
- GroupB (Conventional AFL PDT group ) (Active Comparator): Group B was treated with conventional AFL-PDT
  Interventions: Drug: Placebo cream application; Drug: lidocaine/prilocaine (5%) application; Device: 2940-nm Er:YAG AFL pretreatment; Drug: MAL application; Other: Measurements of the fluorescence intensity; Device: irradiation with red light-emitting diode lamp

INTERVENTIONS:
Drug: Topical Vitamin D (Calcipotriol) application — Calcipotriol ointment 50 mcg/g (Daivonex, Leo Pharma, Denmark) was applied twice for daily on treatment area for 15 consecutive days.
  Arms: GroupA (Vit-D pretreated AFL-PDT group )
Drug: Placebo cream application — placebo cream (indistinguishable from calcipotriol cream by visual and physical appearance and sense of smell) was applied twice for daily on treatment area for 15 consecutive days.
  Arms: GroupB (Conventional AFL PDT group )
Drug: lidocaine/prilocaine (5%) application — For AFL pre-treatment, lidocaine/prilocaine (5%) cream (EMLA; Astra Pharmaceuticals, LP, Westborough, MA, USA) was applied to the treatment area under occlusion for 30 min
Device: 2940-nm Er:YAG AFL pretreatment — After the anaesthetic cream was removed, AFL therapy was performed using a 2940-nm Er:YAG AFL (Joule; Sciton Inc., Palo Alto, CA, USA) at 300-550 µm ablation depth, level 1 coagulation, 22% treatment density and a single pulse
Drug: MAL application — Immediately after AFL treatment, an approximately 1- mm-thick layer of MAL (Metvix, PhotoCure ASA, Oslo, Norway) was applied to the lesion and on 5 mm of surrounding normal tissue. Incubation time is 3 hours
Other: Measurements of the fluorescence intensity — After 3 hours of application with MAL, saline wash was performed and fluorescence imaging analysis was performed with ultraviolet examination light (model 31602,356 nm; Burton Medical Products Crop.) at 10 cm height above the base of each lesion. The red fluorescence (610 nm-700 nm) was separated and extracted by ImageJ program and then used to measure the amount of 633 nm fluorescence of protoporphyrin IX.
Device: irradiation with red light-emitting diode lamp — After incubation for 3 hours, the dressing and cream were removed, and the area was cleansed with saline. The area was irradiated with a red light-emitting diode lamp (Aktilite CL 128; PhotoCure ASA, Oslo, Norway) with peak emission at 632 nm, placed 5 cm away from the skin surface, and a total light dose of 37 J/cm-2. All patients wore protective goggles during illumination.

SUMMARY:
Vitamin D(Vit D) is a pro-differentiation agent that enhances the accumulation of protoporphyrin IX (PpIX) after MAL(methyl-aminolevulinate) incubation in actinic keratosis and may have significant benefit for the treatment of actinic keratosis by ablative fractional laser-primed photodynamic therapy (AFL-PDT).

DETAILED DESCRIPTION:
Photodynamic therapy (PDT) with methyl-aminolevulinate (MAL) is effective in the treatment of actinic keratosis (AK). Many strategies have been studied to improve the production of protoporphyrin IX (PpIX), to improve efficacy of PDT. Pre-treatment of the skin with fractional laser resurfacing is a novel alternative technique to improve the efficacy of PDT for AK. The investigators' previous studies showed that ablative fractional laser primed PDT (AFL-PDT) offered higher efficacy than conventional MAL-PDT in the treatment of AK. But, reduced response rates are also observed in thicker skin lesions, which may be due to insufficient PpIX accumulation within the target tissue.

Cellular differentiation leads to increased synthesis of PpIX from MAL and consecutively, differentiation therapy enhances photosensitization effect. Topical calcipotriol is a well-known pro-differentiation hormone and was demonstrated to influence the effect of PDT on keratinocytes.

The aim of this study was to evaluate efficacy of topical vitamin D in AFL-PDT for AK treatment. Consequently, the investigator compared efficacy, recurrence rate, cosmetic outcome and safety between VitD - AFL-PDT and conventional AFL-PDT.

ELIGIBILITY:
Inclusion Criteria:

* Korean patients aged ≥ 18 years who had biopsy-confirmed Actinic keratosis lesions

Exclusion Criteria:

* calcium metabolic disorder patients
* photosensitivity disorder patients
* lactating or pregnant women
* patients with porphyria or a known allergy to any of the constituents of the MAL cream and lidocaine
* patients with systemic disease, history of malignant melanoma, tendency of melasma development or keloid formation, any AK treatment of the area in the previous 4 weeks, or any conditions associated with a risk of poor protocol compliance; and patients on immunosuppressive treatment

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Differences of short-term complete response rates between VitD-AFL-PDT and AFL-PDT | Short-term complete response rates were evaluated at 3 months after treatment
  Lesion responses were classified as either a complete response (complete disappearance of the lesion) or a noncomplete response (incomplete disappearance)
Differences of long-term complete response rates between VitD-AFL-PDT and AFL-PDT | Long-term complete response rates were evaluated at 12 months
  In all cases of complete response, the patients were reviewed at 12 months to check for recurrence. Recurrence was assessed by inspection, dermoscopy, photography, palpation, and histologic findings. For the histopathologic evaluation of treatment response, at the 12-month follow-up visit, a 3-mm punch biopsy of the treated AK lesion was performed in all cases of clinically incomplete response.
Difference of the recurrence rates between VitD-AFL-PDT and AFL-PDT | Recurrence rates were evaluated respectively at 12 months after treatment.
  In all cases of complete response, the patients were reviewed at 12 months to check for recurrence. Recurrence was assessed by inspection, dermoscopy, photography, palpation, and histologic findings. For the histopathologic evaluation of treatment response, at the 12-month follow-up visit, a 3-mm punch biopsy of the treated AK lesion was performed in all cases of clinically incomplete response.

SECONDARY OUTCOMES:
Differences of cosmetic outcomes between VitD-AFL-PDT and AFL-PDT | The overall cosmetic outcome was assessed 12 months after treatment
  Cosmetic outcomes were graded as excellent (slight redness or pigmentation change), good (moderate redness or pigmentation change), fair (slight-to-moderate scarring, atrophy, or induration), or poor (extensive scarring, atrophy, or induration)
Difference of adverse events (erythema, post-inflammatory hyperpigmentation, edema, itching, oozing, bleeding) rates between VitD-AFL-PDT and AFL-PDT | Within 12 months after each treatment
  Adverse events reported by the patient were noted at each follow-up visit, including severity, duration and need for additional therapy. All events due to PDT were described as phototoxic reactions (i.e., erythema, post-inflammatory hyperpigmentation, oedema, itching, oozing, bleeding and so forth).

OTHER OUTCOMES:
Differences of the fluorescence intensity between VitD-AFL-PDT and AFL-PDT | After 3 hours of application with MAL, fluorescence intensity imaging was assessed 10 minutes before illumination.
  After 3 hours of application with MAL, Fluorescence imaging analysis was performed on treatment area with ultraviolet examination light (model 31602,356 nm; Burton Medical Products Crop.) at 10 cm height above the base of each lesion. The red fluorescence was separated and extracted by ImageJ program and then used to measure the amount of 633 nm fluorescence of protoporphyrin IX.

CONTACTS AND LOCATIONS:
Locations (1):
- Dong-A University, Busan, Seo-gu, Korea, Republic Of, 602-715, South Korea

IPD SHARING:
Plan to Share IPD: No